CLINICAL TRIAL: NCT03843385
Title: Longterm Transfer of FRozen Encapsulated Multidonor Stool Filtrate or Encapsulated Multidonor Microbiome for Chronic Active Ulcerative COlitis
Brief Title: Transfer of FRozen Encapsulated Multidonor Stool Filtrate for Active Ulcerative COlitis
Acronym: FRESCO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Andreas Stallmach (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor-Investigator, Andreas Stallmach, coordinating investigator, Jena University Hospital
Organization: Jena University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KS2017-114
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Diseases
Keywords: fecal transplantation; multidonor fecal transplantation
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive intensive dosing multi-donor FMFT or FMT as therapeutic strategies or saline as a placebo comparator. To achieve balanced distributions for pretreatment factors, we propose to apply stratified (stratum 1: "biologicals yes/no"; stratum 2: "participating centre") block randomization.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To address "concealment of allocation", the randomization will be done centrally and each patient who is randomized and who received one of the compared treatments is part of the full analysis set (ITT analysis set).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- faecal microbiota filtrate (Experimental): Encapsulated faecal microbiota filtrate . 2×5 frozen capsules by mouth on 5 consecutive days per week (5 days on and 2 days off; week 1 - week 12) with water or cool drink.
  Interventions: Drug: encapsulated faecal microbiota filtrate
- faecal microbiota (Active Comparator): Encapsulated faecal microbiota. 2×5 frozen capsules by mouth on 5 consecutive days per week (5 days on and 2 days off; week 1 - week 12) with water or cool drink.
  Interventions: Drug: encapsulated faecal microbiota
- Placebo (Sham Comparator): Placebo: Encapsulated sterile saline. 2×5 frozen capsules by mouth on 5 consecutive days per week (5 days on and 2 days off; week 1 - week 12) with water or cool drink.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: encapsulated faecal microbiota filtrate — Multidonor stool mixed with sterile normal saline, homogenized, filtered, centrifuged, air pressure filtered, encapsulated in hypromellose capsules and frozen.
  Other Names: FMFT
  Arms: faecal microbiota filtrate
Drug: encapsulated faecal microbiota — Multidonor stool mixed with sterile normal saline, homogenized, filtered, encapsulated in hypromellose capsules and frozen.
  Other Names: FMT
  Arms: faecal microbiota
Drug: Placebo — Sterile saline encapsulated in hypromellose capsules and frozen.
  Other Names: Encapsulated sterile saline
  Arms: Placebo

SUMMARY:
FRESCO is a randomized, longitudinal, prospective, three arm, multicentre, double blind study to determine safety and efficacy of repeated faecal microbiota transplantation (FMT) or faecal microbiota filtrate transplantation (FMFT) compared to placebo using oral, frozen capsules in 174 randomized patients with mild to moderate active Ulcerative Colitis.

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a chronic inflammatory bowel disease with significant morbidity and mortality. Although the precise cause remains unknown, disturbances in the intestinal microbial community and changes in the crosstalk between the microbiota and the mucosal immune system have been linked to its pathogenesis. As current therapies are limited, there is a medical need for new therapies. Faecal microbiota transplantation (FMT) has been proven to be effective in managing relapsing Clostridium difficile infection (CDI) and preliminary results indicated that also the transfer of filtrates of donor stool (FMFT) drives gastrointestinal microbiota changes and eliminate symptoms in CDI patients. FRESCO is a randomized, longitudinal, prospective, three arm, multicentre, double blind study to determine safety and efficacy of repeated FMT or FMFT compared to placebo using oral, frozen capsules in 174 randomized patients with mild to moderate active UC. The primary outcome will be clinical and endoscopic remission at week 12. This proposal aims to examine: (a) the efficacy of FMT / FMFT as a therapy for active UC, (b) the safety of FMT / FMFT in patients with UC and (c) the microbial and inflammable changes that occur after FMT / FMFT, to help understand how and why it works in this group of patients. All analyses will be conducted in both intention-to-treat (primary) and per-protocol (sensitivity analyses) populations, and the differences in remission rates and relapse rates between the groups will be statistically analysed to determine the efficiency of FMT versus FMFT.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Prior endoscopic confirmation of UC of at least 6 months AND with a minimum disease extent of 15 cm from the anal verge.
* Having active disease, defined with a Mayo Score between 4-10 and Mayo endoscopic subscore >1
* Failure of conventional therapy or treatment with biologicals and / or small molecules.
* previous medical therapy:

  * oral 5-ASA compounds (5-ASA); stable dosing for 4 weeks before randomization;
  * Azathioprine, 6-Mercaptopurine (6-MP) or Methotrexate (MTX); stable dosing for 8 weeks before randomization;
  * Oral corticosteroid therapy (prednisone ≤ 20 mg/day or budesonide ≤ 9 mg/day); stable dosing for 2 weeks before randomization;
  * Topical therapy (foams, clysms) with mesalazine or budesonide: stable dosing for 2 weeks before randomization.
* previous vaccination against SARS-CoV-2 or previous SARS-CoV-2 infection or positive serology
* Ability to understand and willingness to sign informed consent document in patients whom the investigator believes can and will comply with the requirements of the protocol.
* Potentially childbearing patient: negative pregnancy test and use of a highly effective contraceptive method

Exclusion Criteria:

* Crohn's disease or indeterminate colitis or proctitis ulcerosa alone
* Acute abdomen or other clinical emergencies (e.g. toxic megacolon, fulminant gastrointestinal hemorrhage, ileus, perforation, etc.)
* Previous operations on the colon: colectomy, partial colon resections
* current gastrointestinal infections
* Congenital or acquired immunodeficiency
* severe comorbidity (e.g. insulin-dependent diabetes mellitus, decompensated liver cirrhosis, primary sclerosing cholangitis, renal impairment > grade 2)
* diagnosis of a malignoma in the last 3 years
* refusal of endoscopies with video documentation
* No specific therapy for ulcerative colitis to date
* Lack of immunity to SARS-CoV-2
* Previous treatment with TNF-, IL12/IL23-, IL23- or integrin-antibodies within the last 8 weeks before randomisation
* Treatment with calcineurin inhibitors within the last 4 weeks before randomization
* Treatment with JAK inhibitors (e.g., tofacitinib, filgotinib, or upadacitinib) within the last 4 weeks prior to randomization
* Treatment with S1P receptor modulators (e.g. ozanimod, etrasimod) within the last 4 weeks before randomization
* Systemic antibiotic treatment within the last 8 weeks prior to randomization.
* Known intolerance of metronidazole or vancomycin
* Previous FMT or FMFT, previous participation in this study (screening allowed)
* Participation in a clinical trial within the last 3 months
* Use of probiotics in tablet, capsule, or powder form, or appropriate drinking yogurts (or similar) within 2 weeks prior to randomization
* Failure to ensure frozen storage of investigational products
* Addictive or other medical conditions or circumstances that do not allow the subject to appreciate the nature, significance, scope, and possible consequences of the clinical trial
* Indications that the patient would be unlikely to comply with the protocol (e.g., unwillingness to cooperate - compliance questionable)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
clinical remission | 12 weeks
  The primary outcome will be clinical remission at week 12 post first transfer of FMFT or FMT, defined by Mayo score ≤ 2, all subscores ≤ 1; additionally patients unavailable at the week 12 follow-up will be included as non-responders (i.e. counted no remission).

SECONDARY OUTCOMES:
steroid-free clinical remission | 12 weeks
  steroid-free clinical remission at week 12 post first transfer of FMFT or FMT, with a minimum of steroid free time of 4 weeks (week 8 to 12)
clinical response | 12 weeks
  clinical response is defined by decrease in partial Mayo score by more than 3 points and a minimum decrease of 30% from output value and additional bleeding subscore by more than 1 point or absolute sub-score of 0-1
change in quality of life | 52 weeks
  quality of life is assessed at week 0,4,8,12 for short-term efficacy and for long-term efficacy at week 24,36 and 52 post first transfer by Inflammatory Bowel Disease Quality of Life Questionnaire (IBDQ). The IBDQ is a 32-item self-rated questionnaire with 4 domains (bowel symptoms, emotional function, social function, systemic symptoms). Each item is rated on a seven-point Likert Scale. The total score ranges from 32 to 224 points with higher scores reflecting better well-being.
endoscopic remission | 12 weeks
  endoscopic remission at week 12 post first transfer of FMFT or FMT, with a score between 0 and 3, (0 = Normal or inactive disease, 1 = mild inflammatory activity, 2 = moderate disease, 3 = severe disease)
mucosal inflammation - measured through fecal calprotectin | 52 weeks
  mucosal inflammation in stool samples at week 0, 4, 8, 12, 24, 36, 52 post first transfer of FMFT or FMT
microbiome analysis | 52 weeks
  analysis of stool samples at week 0, 4, 8, 12, 24, 36, 52 post first transfer of FMFT or FMT regarding microbiome diversity and composition
virome analysis | 52 weeks
  analysis of stool samples at week 0, 4, 8, 12, 24, 36, 52 post first transfer of FMFT or FMT regarding virome composition
MAYO Total Score | 52 weeks
  Comparison of the MAYO total Score between the 3 Arms (FMFT, FMT and Placebo)
Histological mucosal inflammation - Nancy index | 12 weeks
  Analysis of obtained mucosa biopsies at week 0 and 12, regarding disease activity graded with the Nancy index
Safety - adverse events and severe adverse events | 52 weeks
  adverse events and severe adverse events in the different treatment arms will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Stallmach, Prof., Study Director — Jena University Hospital
Locations (15):
- Germany (15):
  - Jena University Hospital, Jena, Thuringia
  - Sozialstiftung Bamberg, Bamberg
  - Charité Berlin, Berlin
  - DRK Kliniken Berlin Westend, Berlin
  - Krankenhaus Waldfriede, Berlin
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - FAU Universität Erlangen-Nürnberg, Erlangen
  - Agaplesion Markus Krankenhaus, Frankfurt
  - Universitätsklinik Freiburg, Freiburg im Breisgau
  - Klinikum Fulda, Fulda
  - Universitätsklinikum Halle (Saale), Halle
  - Universitätsklinikum Schleswig Holstein, Kiel
  - Gesellschaft Klinische Studien Leipzig, Leipzig
  - Städtisches Klinikum Lüneburg, Lüneburg
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stallmach A, Grunert P, Stallhofer J, Loffler B, Baier M, Rodel J, Kiehntopf M, Neugebauer S, Pieper DH, Junca H, Tannapfel A, Merkel U, Schumacher U, Breternitz-Gruhne M, Heller T, Schauer A, Hartmann M, Steube A. Transfer of FRozen Encapsulated multi-donor Stool filtrate for active ulcerative Colitis (FRESCO): study protocol for a prospective, multicenter, double-blind, randomized, controlled trial. Trials. 2022 Feb 22;23(1):173. doi: 10.1186/s13063-022-06095-1. PMID 35193638